CLINICAL TRIAL: NCT02274753
Title: Personalizing Colorectal Cancer Medicine: an Integrative Approach for the Identification of Prognostic Parameter Combinations at the Time of Surgery and During the Follow-up
Brief Title: Personalizing Colorectal Cancer Medicine (ImmuCol2)
Acronym: ImmuCol2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: NI13017
Record Dates: First submitted 2014-10-20; First posted 2014-10-24 (Estimated); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The pathologist of each center will choose a tumor block containing the core of the tumor and the invasive margin. Seven tissues sections (five of 4 microns and two of 20 microns) of this tumor bmock will be cut and deposited on glass slides for the immunohistochemical and tumor genetic analysis. If biopsies for diagnostic purpose are available in the laboratory of pathology for the same patient, two tissue sections of 4 microns of each biopsy will be cut and deposited on a glass slide. Two tubes of blood (5 ml tube without anticoagulant) and a 10 ml tube with EDTA will be taken in consultation or hospitalization before the first chemotherapy and at 1 year, 2 years and 3 years. These samples will be used for gene expression analysis and in the search for biological signs of autoimmunity.
Oversight: Data Monitoring Committee: No

SUMMARY:
Colorectal cancers are the leading cancers for both sexes combined. They represent 15-20% of all cancers. This cancer has a severe prognosis, the survival rate at 5 years is around 55% and in France it is estimated, all colorectal cancers are responsible for an annual mortality of 15,000 patients. The prognosis of colon cancer knows no significant improvement.

The treatment of colon cancer is surgical. It is intended for removal of colonic segment bearing the tumor with margins of healthy colon. The therapeutic attitude following the surgery is essentially driven by histopathology of the tumor. Adjuvant chemotherapy for all patients with localized stage II provides no benefit because the effectiveness of chemotherapy is limited and vulnerable to systemic toxicity. However, nearly 30% of patients with stage II disease will have a recurrence / metastasis. These patients could benefit from adjuvant chemotherapy.

Intense research efforts have been made to identify markers predictive of relapse. Over thirty biological markers (eg. Mutations, deletions, chromosomal instability, ...) were highlighted. None of them has so far sufficient prognostic value (independent of TNM) to justify routine application in clinical practice in order to adapt the treatment of patients.

The identification of new prognostic markers is a major issue for colorectal cancer. We showed that the intratumoral density memory T lymphocytes (CD45RO) and cytotoxic (CD8) strongly influenced the clinical outcome of patients. We have developed and validated a "immunoscore" technique intratumoral immune quantification and creates a platform to facilitate the clinical immuno transfer.

We are currently conducting a large international retrospective study (22 centers,> 9000 patients) with promotion of cancer immunotherapy Company (SITC) to validate the method "immunoscore." At the same time, we are conducting a prospective multicenter study "ImmuCol" (National PHRC) to validate the prognostic value of "immunoscore" in colorectal cancer stage I-IV. The goal of inclusion has been achieved, as 420 patients were included for 18 months. Clinical follow-up will be 3 years after surgery.

The program ImmuCol2 research takes advantage of the ImmuCol study to extend the investigation beyond the immunoscore to define the combination of interest, prognostic and theranostic parameters at diagnosis and during the clinical course patients with an objective of personalized medicine.

DETAILED DESCRIPTION:
The project aims:

(i) to combine at time of diagnosis the immunoscore with parameters related to the patient, its tumor and the associated microenvironment (ii) to detect events occurring during the follow up period that could modify the initial prognosis and lead to a repositioning of the patient, to move towards a dynamic personalized medicine.

(iii) to explore the Theranostic aspect of the parameters monitored at the time of diagnosis for patients with colonic cancers treated with adjuvant chemotherapy.

To this end we will investigate:

* Tumor's features:

  - We will determine the microsatellite instability status and search for mutations of 46 genes (ABL1, AKT1, ALK, APC, ATM, BRAF, CCDH1, CDKN2A, CSF1R, CTNNB, EGFR, ERBB2, ERBB4, EZH2, FBXW7, FGFR1, FGFR2, FGFR3, FLT3, GNA11, GNAQ, GNAS, HNF1A, HRAS, IDH1, IDH2, JAK2, JAK3, KDR, KIT, KRAS, NOTCH1, NPM1, NRAS, PDGFRA, PDGFRA, PIK3CA, PTEN, PTPN11, RB1, RET, SMAD4, SMARCB1, SMO, STK11, TP53, VHL) by next generation sequencing (NGS).
* Tumor immune microenvironment features:

  - 24 immune related genes, 24 miRNA and co-inihibitory molecules (PD1, PD1-L, LAG-3, TIM3, CTLA-4) will be explored on tumor samples.
* Systemic disorders:

  * Autoimmunity, allergy or inflammatory diseases will be sought with a dedicated questionnaire filled out by the patient and a serum examination for the screening of immune disorders at the time of diagnosis and during the survey.
  * The nutritional status (% of weight loss) and the deficiencies in vitamins, folic acid, trace elements and thyroid hormones that synergise with immune cells will be determined at the time of diagnosis.
* Psychological status:

  - The impact of the psychological profile of the patient will be investigated with a dedicated questionnaire, given at the time of diagnosis and every six months.
* Data mining to achieve a dynamic personalized medicine:

The integration and statistical analysis of heterogeneous data types (clinical and different experimental data) will be performed using with tranSMART, an open source platform and with bioinformatic tools (TMEdb, ClueGO, CluePedia, Genesis) developed by participant teams.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with newly diagnosed colon cancer
* Patient with signed informed consent
* Patient follow-up during the first three years made in the recruiting center

Exclusion Criteria:

* Adjuvant treatment (chemotherapy) started at the time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with newly diagnosed colon cancer.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2015-03-11 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Relapse in relation with the immunoscore determined on a tumor section and criteria defined in the monitoring of patients | 3 years
  This primary outcome (relapse) will be correlated to the immunoscore and several criteria (dysimmune systemic criteria, malnutrition, vitamin deficiencies in micronutrients, psychological criteria) in order to evaluate their pronostic impact. The measure is a composite outcome.

SECONDARY OUTCOMES:
Relapse in relation with the immune component cancers beyond immunoscore | Every 3 months during 2 years and every 6 months during the third year
  The primary outcome (relapse) will be correlated to the expression of immune molecules associated with activation or inhibition of T lymphocyte and by in situ analysis of the expression level of immune genes. A comparison of the prognostic performance of these parameters will be performed. These parameters will then be analyzed in combination with immunoscore to determine the optimal combination of immune parameters with prognostic and theranostic target.
Relapse in relation with the immunoscore on biopsies | Every 3 months during 2 years and every 6 months during the third year
  The primary outcome (relapse) will be correlated to the immunoscore and expression of immune genes determined on biopsies performed for diagnosis purpose

CONTACTS AND LOCATIONS:
Overall Officials: Franck Pages, Professor (MD-PHD), Principal Investigator — AP-HP; Paris Descartes University
Locations (9):
- France (9):
  - Hopital de Besançon (CHU), Besançon
  - Hopital Avicenne, Bobigny
  - CHU de Bordeaux, Bordeaux
  - Institut Bergonié Bordeaux, Bordeaux
  - Hopital Beaujon, Clichy
  - Hopital de Dijon (CHU), Dijon
  - Hopital Europeen Georges Pompidou (HEGP), Paris
  - Hopital de Poitiers (CHU), Poitiers
  - Hopital Charles Nicolle (CHU), Rouen

REFERENCES:
- [Background] Dunn GP, Bruce AT, Ikeda H, Old LJ, Schreiber RD. Cancer immunoediting: from immunosurveillance to tumor escape. Nat Immunol. 2002 Nov;3(11):991-8. doi: 10.1038/ni1102-991. PMID 12407406
- [Background] Saltz LB, Kelsen DP. Adjuvant treatment of colorectal cancer. Annu Rev Med. 1997;48:191-202. doi: 10.1146/annurev.med.48.1.191. PMID 9046955
- [Background] Pages F, Berger A, Camus M, Sanchez-Cabo F, Costes A, Molidor R, Mlecnik B, Kirilovsky A, Nilsson M, Damotte D, Meatchi T, Bruneval P, Cugnenc PH, Trajanoski Z, Fridman WH, Galon J. Effector memory T cells, early metastasis, and survival in colorectal cancer. N Engl J Med. 2005 Dec 22;353(25):2654-66. doi: 10.1056/NEJMoa051424. PMID 16371631
- [Background] Galon J, Costes A, Sanchez-Cabo F, Kirilovsky A, Mlecnik B, Lagorce-Pages C, Tosolini M, Camus M, Berger A, Wind P, Zinzindohoue F, Bruneval P, Cugnenc PH, Trajanoski Z, Fridman WH, Pages F. Type, density, and location of immune cells within human colorectal tumors predict clinical outcome. Science. 2006 Sep 29;313(5795):1960-4. doi: 10.1126/science.1129139. PMID 17008531
- [Background] Pages F, Kirilovsky A, Mlecnik B, Asslaber M, Tosolini M, Bindea G, Lagorce C, Wind P, Marliot F, Bruneval P, Zatloukal K, Trajanoski Z, Berger A, Fridman WH, Galon J. In situ cytotoxic and memory T cells predict outcome in patients with early-stage colorectal cancer. J Clin Oncol. 2009 Dec 10;27(35):5944-51. doi: 10.1200/JCO.2008.19.6147. Epub 2009 Oct 26. PMID 19858404
- [Background] Mlecnik B, Tosolini M, Kirilovsky A, Berger A, Bindea G, Meatchi T, Bruneval P, Trajanoski Z, Fridman WH, Pages F, Galon J. Histopathologic-based prognostic factors of colorectal cancers are associated with the state of the local immune reaction. J Clin Oncol. 2011 Feb 20;29(6):610-8. doi: 10.1200/JCO.2010.30.5425. Epub 2011 Jan 18. PMID 21245428
- [Background] Galon J, Mlecnik B, Bindea G, Angell HK, Berger A, Lagorce C, Lugli A, Zlobec I, Hartmann A, Bifulco C, Nagtegaal ID, Palmqvist R, Masucci GV, Botti G, Tatangelo F, Delrio P, Maio M, Laghi L, Grizzi F, Asslaber M, D'Arrigo C, Vidal-Vanaclocha F, Zavadova E, Chouchane L, Ohashi PS, Hafezi-Bakhtiari S, Wouters BG, Roehrl M, Nguyen L, Kawakami Y, Hazama S, Okuno K, Ogino S, Gibbs P, Waring P, Sato N, Torigoe T, Itoh K, Patel PS, Shukla SN, Wang Y, Kopetz S, Sinicrope FA, Scripcariu V, Ascierto PA, Marincola FM, Fox BA, Pages F. Towards the introduction of the 'Immunoscore' in the classification of malignant tumours. J Pathol. 2014 Jan;232(2):199-209. doi: 10.1002/path.4287. PMID 24122236
- [Background] Myron Kauffman H, McBride MA, Cherikh WS, Spain PC, Marks WH, Roza AM. Transplant tumor registry: donor related malignancies. Transplantation. 2002 Aug 15;74(3):358-62. doi: 10.1097/00007890-200208150-00011. PMID 12177614
- [Background] Dalerba P, Maccalli C, Casati C, Castelli C, Parmiani G. Immunology and immunotherapy of colorectal cancer. Crit Rev Oncol Hematol. 2003 Apr;46(1):33-57. doi: 10.1016/s1040-8428(02)00159-2. PMID 12672517
- [Background] Jass JR. Lymphocytic infiltration and survival in rectal cancer. J Clin Pathol. 1986 Jun;39(6):585-9. doi: 10.1136/jcp.39.6.585. PMID 3722412
- [Background] Phillips SM, Banerjea A, Feakins R, Li SR, Bustin SA, Dorudi S. Tumour-infiltrating lymphocytes in colorectal cancer with microsatellite instability are activated and cytotoxic. Br J Surg. 2004 Apr;91(4):469-75. doi: 10.1002/bjs.4472. PMID 15048750
- [Background] Pages F, Galon J, Dieu-Nosjean MC, Tartour E, Sautes-Fridman C, Fridman WH. Immune infiltration in human tumors: a prognostic factor that should not be ignored. Oncogene. 2010 Feb 25;29(8):1093-102. doi: 10.1038/onc.2009.416. Epub 2009 Nov 30. PMID 19946335
- [Background] Fridman WH, Pages F, Sautes-Fridman C, Galon J. The immune contexture in human tumours: impact on clinical outcome. Nat Rev Cancer. 2012 Mar 15;12(4):298-306. doi: 10.1038/nrc3245. PMID 22419253
- [Background] Bindea G, Mlecnik B, Tosolini M, Kirilovsky A, Waldner M, Obenauf AC, Angell H, Fredriksen T, Lafontaine L, Berger A, Bruneval P, Fridman WH, Becker C, Pages F, Speicher MR, Trajanoski Z, Galon J. Spatiotemporal dynamics of intratumoral immune cells reveal the immune landscape in human cancer. Immunity. 2013 Oct 17;39(4):782-95. doi: 10.1016/j.immuni.2013.10.003. PMID 24138885